CLINICAL TRIAL: NCT07195136
Title: Investigation of the Effect of Orange Blossom Essential Oil Placed in the Stoma Bag on Odor Removal, Social Isolation, and Stoma Adaptation in Individuals With Stoma
Brief Title: Orenage Blossom Oil Essential Application in Stoma
Acronym: Stoma Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Meltem Akbaş, Dr, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 06.09.2024/145; Cukurova University (Other: Cukurova University)
Record Dates: First submitted 2025-09-17; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Stoma; Nursing; Nursing Care; Essential Oil
Keywords: stoma; nursing; nursin care; essenntial oil
MeSH Terms: interventions — Oils, Volatile

STUDY DESIGN:
Intervention Model Description: Using the Training Brochure, participants were instructed, lasting approximately 15 minutes, to place 10 drops of orange blossom essential oil into their clean bags during colostomy bag changes and spread the oil throughout the entire inner surface of the bag. During this training, the application was first administered by the researcher, and then performed by the patient under the researcher's supervision. The patients in the experimental group were provided with orange blossom essential oil by the researcher for use for one month.
Who Masked: Participant
Masking Description: Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): essential oil
  Interventions: Behavioral: Essential Oil
- control (No Intervention): standart care

INTERVENTIONS:
Behavioral: Essential Oil — essential oil
  Arms: intervention

SUMMARY:
Because the stoma will become a part of the individual's body and directly impact their quality of life, careful attention should be paid to its location and surgical procedure. Stoma care nurses should provide effective training to patients and those responsible for their care. Patients and their families should be regularly monitored, followed up, and cared for at home after discharge. They should also be provided with information about appropriate units to consult if any problems arise. Stoma support groups should be established to foster social interaction. A well-planned surgical procedure protects individuals from the development of complications and problems that can be considered a "life sentence."

DETAILED DESCRIPTION:
This prospective, randomized, controlled study aims to investigate the effects of orange blossom essential oil placed in the stoma bag on odor reduction, social isolation, and stoma compliance in individuals with permanent colostomies. Sample size calculations were performed using a priori power analysis (t-test) for the intervention and control groups. Accordingly, with an effect size of d=1.12, a 5% error rate (α=0.05), and 80% power (1-β=0.80), the minimum sample size for both groups was calculated as 54. Considering potential losses, the total sample size will be increased by 10%, with 30 patients in each group (Experimental Group: 30, Control Group: 30), for a total of 60 patients. Data will be collected using a patient personal information form, a patient information form, a compliance scale for individuals with stoma, and a social isolation scale, all prepared by the researchers based on literature.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Over 18 years of age
* With a stoma
* No stoma-related complications

Exclusion Criteria:

* Leaving the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Stoma Adaptation Scale | 30 day
  Scale items are scored between 0 and 4. The minimum score is 0 and the maximum is 92. A higher score indicates greater compliance with the stoma.
Social Isolation Scale | 30 day
  Scale items are scored on a 1-3 scale. The minimum score is 14 and the maximum is 42. As the score increases, the level of social isolation increases.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Akbaş, Principal Investigator — Universty Of Cukurova

IPD SHARING:
Plan to Share IPD: No